CLINICAL TRIAL: NCT04203667
Title: Prospective, Multicenter Study for the Evaluation of Safety and Performance of the Interscope EndoRotor Endoscopic Mucosal Resection System for the Removal of Alimentary Tract Mucosa in the Colon
Brief Title: EndoRotor® Endoscopic Mucosal Resection System for the Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interscope, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0001
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Polyp of Colon; Endoscopic Mucosal Resection; Recurrent Colon Adenoma
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Post-market, prospective, non-randomized, multi-center study for the treatment of subjects with the need for resection of recurrent flat or sessile colorectal lesions where EndoRotor is the primary resection modality of persistent adenoma with a scarred base.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EndoRotor Resection Arm (Other): All participants enrolled in this study will undergo treatment with the EndoRotor during colonoscopy for endoscopic mucosal resection in the colon to resect and remove tissue, not intended for biopsy, of the gastrointestinal system including post-endoscopic endoscopic mucosal resection of tissue persistence with a scarred base and residual tissue from peripheral margins following endoscopic mucosal resection.
  Interventions: Device: EndoRotor Resection

INTERVENTIONS:
Device: EndoRotor Resection — The EndoRotor® is a powered cutting cannula for the removal of alimentary tract mucosa. Cutting is performed by aspirating tissue into a rotating cutting window. The resected tissue is immediately aspirated away from the resection site and collected in the EndoRotor Specimen Trap. The tissue can then be sent for pathological examination using standard methods.
  The system consists of a power console, foot control, specimen trap with pre-loaded filter and the applied part, which is the single-use catheter.

SUMMARY:
The EndoRotor® is intended for use (USA labeling) in endoscopic procedures by a trained gastroenterologist to resect and remove tissue, not intended for biopsy, of the gastrointestinal (GI) system including post-endoscopic mucosal resection (EMR) tissue persistence with a scarred base and residual tissue from the peripheral margins following EMR.

In this trial investigators will conduct a post-market, prospective, non-randomized, multi-center study for the treatment of subjects with the need for resection of recurrent flat or sessile colorectal lesions where EndoRotor is the primary resection modality of persistent adenoma with a scarred base.

DETAILED DESCRIPTION:
Although the majority of polyps are non-malignant, it is known that the risk of malignancy increases with polyp size, with polyps < 10 mm having < 1% risk of cancer, polyps of 10 mm having a 10% risk of cancer and polyps of 20 mm having a greater than 10% risk of cancer. It is also understood that a polyp of < 1 cm takes approximately 10 years to transform into invasive colorectal carcinoma. Therefore, adenomas greater than 5 mm are normally treated. Polyps with tethered bases resulting from scarring are often the most challenging to resect endoscopically. The scarring can be caused by previous attempts at resection, previous deep biopsies, or tattoos placed too closely. These polyps often do not lift and can be impossible to snare even when stiff snares are used. Endoscopic submucosal dissection (ESD) and knife-assisted resection (KAR) are techniques that have been shown effective in the management of scarred polyps, however these techniques have not been widely adopted in the West. Argon plasma coagulation has been more commonly used to ablate adenomatous tissue in scarred polyps but this technique does not allow for the histological assessment of the scarred polyp and is less effective than ESD. The EndoRotor provides a technique whereby the lesion can be effectively removed without adjunct procedures with collection of tissue for histological assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥18 to ≤85 years.
2. At least one recurrent flat or sessile colorectal lesion measuring up to 6 cm in diameter and/or length.
3. Presence of recurrent flat or sessile lesion where the EndoRotor may be used to resect recurrent neoplasia.
4. Favorable anatomy that allows the investigator to access the lesion.
5. Subject is able and willing to comply with site standard medical follow-up, including the 90-day follow-up visit.
6. Subject has been informed of the nature of the study, agrees to participate and has signed the consent form.

Exclusion Criteria:

1. Inability to give informed consent.
2. Subject age is <18 years of age or >85 years of age.
3. Presence of a lesion that represents cancer or has a high chance of harboring submucosal invasive cancer.
4. Presence of synchronous lesions intended for resection that would require use of a concomitant resection modality
5. Medical reasons the procedure cannot be performed (i.e. labile blood pressure, anticoagulation laboratory levels that are too high and risk excessive bleeding, systemic infection, etc.)
6. Active antiplatelet therapy (Plavix , 325mg aspirin therapy) - patient off treatment for < 1 week.
7. Inability to undergo a procedure under propofol sedation or General Anesthesia.
8. Female patients who are known to be pregnant.
9. Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g., severe chronic obstructive pulmonary disease, hepatic failure, cardiac disease, autoimmune disorders or conditions of severe immunosuppression).
10. Any clinical evidence that the investigator feels would place the subject at increased risk with the deployment of the device.
11. Subject is participating in another study of a device, medication, biologic, or other agent within 90 days and could, in the opinion of the investigator, impact the results of this study.
12. Subject has other medical, social or psychological problems that in the opinion of the investigator would preclude them from receiving this treatment and the procedures and participating in evaluations pre- and post-treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, MD, Principal Investigator — Principal Investigator
Locations (11):
- Geisinger Medical Center, Danville, Pennsylvania, United States
- France (3):
  - Centre Hospitalier Universitaire (CHU), Angers
  - Hopital Edouard Herriot, Lyon
  - Cochin University Hospital, Paris
- Germany (4):
  - Allgemeines Krankenhaus Celle, Celle
  - Clinic and Polyclinic for Interdisciplinary Endoscopy University Hospital Hamburg Eppendorf, Hamburg
  - Catholic Clinic Mainz, Mainz
  - Sana Klinikum Offenbach, Offenbach
- Italy (3):
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Università Cattolica del Sacro Cuore, Instituto di Clinica Chirurgica, Rome
  - Humanitas Research Hospital & Humanitas University, Rozzano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knabe M, Maselli R, Cesbron-Metivier E, Hollerbach S, Petruzziello L, Prat F, Khara HS, Pioche M, Hartmann D, Cesaro P, Barbaro F, Berger A, Spada C, Diehl DL, May A, Ponchon T, Repici A, Costamagna G. Endoscopic powered resection device for residual colonic lesions: the first multicenter, prospective, international clinical study. Gastrointest Endosc. 2024 May;99(5):778-786. doi: 10.1016/j.gie.2023.11.050. Epub 2023 Dec 1. PMID 38042207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 12 centers in the US and Europe. First participant was enrolled in the study on January 25, 2018 and the last participant was enrolled in the study on June 24, 2020.
  Of the 80 patients screened for this study, 66 were enrolled and treated with EndoRotor.
Pre-assignment Details: The study was over-enrolled. The protocol required 60 subjects; however, 66 subjects were enrolled and treated of which 62 completed the study.
Groups:
- EndoRotor Resection Arm: All participants enrolled in this study will undergo treatment with the EndoRotor during colonoscopy for endoscopic mucosal resection in the colon to resect and remove tissue, not intended for biopsy, of the gastrointestinal system including post-endoscopic endoscopic mucosal resection of tissue persistence with a scarred base and residual tissue from peripheral margins following endoscopic mucosal resection.
  EndoRotor Resection: To collect data in support of the safety and performance of the Interscope EndoRotor® Endoscopic Mucosal Resection System on a post-market basis. The study will confirm that the EndoRotor resections are safe and effective in the removal of recurrent adenoma. post Endoscopic Mucosal Resection.
Period: Overall Study
Arm/Group | EndoRotor Resection Arm
Started (Intent to Treat Population) | 66
Per Protocol Population | 45
Completed | 62
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — PI left center and never scheduled 90 day follow-up visit. | 1

BASELINE CHARACTERISTICS:
Population: Patients who were enrolled in the study.
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 49
  Not Disclosed | 16
  African/Black | 1
Height [Mean (Standard Deviation); unit: cm] | 168.2 (10.0)
Weight [Mean (Standard Deviation); unit: kg] | 76.1 (17.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 135.6 (25.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 76.1 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint Defined as the Ability of the EndoRotor to Resect Lesions Without Concomitant Use of Other Resection Modalities and With no Device-related Serious Adverse Events Through the 90 Day Post Procedure Follow-up Visit.
Time Frame: Index Procedure through 90 Day Post Procedure Follow-up Visit
Population: Primary endpoint analysis will be completed on the per protocol population which consists of subjects who had complete lesion resection with the EndoRotor alone without any adjunctive modality resection, did not have inclusion/exclusion protocol deviations, and completed the 90 day follow-up visit.
Measure: Count of Participants; unit: Participants
Groups:
- EndoRotor Resection Arm: All participants enrolled in this study will undergo treatment with the EndoRotor during colonoscopy for endoscopic mucosal resection in the colon to resect and remove tissue, not intended for biopsy, of the gastrointestinal system including post-endoscopic endoscopic mucosal resection of tissue persistence with a scarred base and residual tissue from peripheral margins following endoscopic mucosal resection.
  EndoRotor Resection: The EndoRotor® is a powered cutting cannula for the removal of alimentary tract mucosa. Cutting is performed by aspirating tissue into a rotating cutting window. The resected tissue is immediately aspirated away from the resection site and collected in the EndoRotor Specimen Trap. The tissue can then be sent for pathological examination using standard methods.
  The system consists of a power console, foot control, specimen trap with pre-loaded filter and the applied part, which is the single-use catheter.
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 45
Participants | 45

2. Primary Outcome: Primary Safety Analysis Defined as the Occurrence of Serious Adverse Events Related to the EndoRotor Device as Measured From the Index Procedure Through the 90 Day Post Procedure Follow-up Visit.
Time Frame: Index Procedure through 90 Day Post Procedure Follow-up Visit
Population: The safety analysis will be completed on all subjects who were treated with the EndoRotor device.
Measure: Number; unit: Serious Adverse Events
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 66
Serious Adverse Events
  Total number of serious adverse events in Intent to Treat Population. | 5
  Delayed Rectal Bleed both mild Relation EndoRotor: probable/possible Relation Proc: Both probable | 2
  Mucosal Laceration Severe Relation to EndoRotor: Unlikely Relation to Procedure: Possible | 1
  Single Arterial Bleed Severe Relation to EndoRotor: Not related Relation to Proc. Not related | 1
  General Infection Moderate Relation to EndoRotor: Not related Relation to Proc. Not related | 1

3. Secondary Outcome: Efficacy Defined as the Number of Participants Where EndoRotor Was Able to Resect the Entire Lesion in a Single Procedure.
Time Frame: Index Procedure
Population: Secondary endpoint analysis will be completed on the per protocol population which consists of subjects who had complete lesion resection with the EndoRotor alone without any adjunctive modality resection, did not have inclusion/exclusion protocol deviations, and completed the 90 day follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 45
Participants | 45

4. Secondary Outcome: Post-resection Stenosis Defined as the Occurrence of Colon Stenosis Following the Index Procedure.
Time Frame: 90-day follow-up visit
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 47
Participants | 0

5. Secondary Outcome: Rate of Disease Persistence Defined as Remnant Disease at the Location of the Index Resection as Determined Endoscopically by the Investigator at the 90 Day Follow-up Visit.
Time Frame: 90-day follow-up visit
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 45
Participants | 21

6. Secondary Outcome: Histologic Assessment Defined as the the Diagnostic Value of the Specimens Collected in the EndoRotor Specimen Trap (Could a Diagnosis be Rendered).
Time Frame: 90-day follow-up visit
Population: as for outcome 3
Measure: Count of Units; unit: Specimens
Units Other Than Participants: Specimens
Arm/Group | EndoRotor Resection Arm
Number analyzed (Participants) | 45
Number analyzed (Specimens) | 45
Specimens | 45

ADVERSE EVENTS:
Time Frame: Index procedure through the 90 day post procedure follow-up visit.
Arm/Group | EndoRotor Resection Arm
All-Cause Mortality (participants affected / at risk) | 1/66
Serious Adverse Events (participants affected / at risk) | 7/66
Other Adverse Events (participants affected / at risk) | 6/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoRotor Resection Arm (N=66)
Mucosal Laceration (Injury, poisoning and procedural complications) | 1 (1) — Onset time: Procedure Severity: Severe Relationship to EndoRotor: Unlikely Relationship to Procedure: Possible Action Taken: Clipping and Hospitalization Outcome: Recovered
Delayed Rectal Bleed (Injury, poisoning and procedural complications) | 2 (2) — Onset: Post Procedure / After Discharge Severity: Mild / Mild Relation EndoRotor: Possible / Probable Relation Procedure: Both Probable Action Taken: Both Hospitalization, observation, no intervention needed Outcome: Both Recovered
Single Arterial Bleed (Gastrointestinal disorders) | 1 (1) — Onset: Procedure Severity: Severe Relationship EndoRotor: Not Related Relationship Procedure: Related Action Taken: clips and hospitalization Outcome: recovered
Delayed Bleeding (Gastrointestinal disorders) | 1 (1) — Onset: post procedure prior to discharge Severity: moderate Relationship to EndoRotor: Not related Relationship to Procedure: Not related Action taken: Mediation, hospitalization, endoscopic hemostasis Recovered
General Infection (Infections and infestations) | 1 (1) — Onset: after discharge prior to 90 day follow-up Severity: moderate Relationship to EndoRotor: Not related Relationship to Procedure: Possible Action taken: Hospitalization and observation Recovered
Urinary Tract Infection (Infections and infestations) | 1 (1) — Onset: After discharge prior to 90 days Severity: Mild Relationship to EndoRotor: Not related Relationship to Procedure: Not related Action taken: Hospitalization Recovered
Heart Attack (Cardiac disorders) | 1 (1) — Onset: After discharge prior to 90 days Severity: Severe Relationship to EndoRotor: Not related Relationship to Procedure: Not related Action taken: None Outcome: Death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoRotor Resection Arm (N=66)
Post Polypectomy Syndrome (Gastrointestinal disorders) | 1 (1) — Onset: post procedure prior to discharge Severity: moderate Relationship to EndoRotor: not related Relationship to procedure: related Action taken: medication Recovered
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) — Onset: Post procedure prior to discharge Severity: mild Relationship to EndoRotor: not related Relationship to Procedure: not related Action: Medication Recovered
Bleeding (Injury, poisoning and procedural complications) | 2 (2) — Onset: Both Procedure Severity: Both mild Relationship to EndoRotor: Possible / Related Relationship to Procedure: Possible / Related Action: Hot biopsy / Clip Both recovered
Seeping bleed (Injury, poisoning and procedural complications) | 2 (2) — Onset: both procedure Severity: both mild Relationship to EndoRotor: both related Relationship to Procedure: both not related Action: both clips Both Recovered

LIMITATIONS AND CAVEATS:
COVID pandemic made follow-up at each center difficult or impossible for patients who had a 90 day follow-up from March 2020 and beyond. Most of Europe was on lockdown from this point through June 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04203667/Prot_SAP_001.pdf